CLINICAL TRIAL: NCT03391622
Title: The Correlation Between Thrombin Generation Values and Percutaneous Coronary Intervention Results in Active Ischemic Heart Disease Patients.
Brief Title: Thrombin Generation Values and Percutaneous Coronary Intervention Results.
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: EMC166-17
Record Dates: First submitted 2017-12-07; First posted 2018-01-05 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Coagulation Disorder; Ischemic Heart Disease; Artery Coronary Stenosis
Keywords: thrombin generation; calibrated automated thrombogram; ischemic heart disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Hemostatic Disorders; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Calibrated Automated Thrombogram — blood samples will be collected . Thrombin generation in platelet-poor plasma will be measured by means of the Calibrated Automated Thrombogram (CAT).

SUMMARY:
Cardiovascular diseases are the most common cause of death in the western world. Myocardial infarction pathogenesis usually involves the development of an atherosclerotic plaque and thrombus.

Past research has shown a correlation between thrombin generation values and ischemic heart disease, however, to our knowledge no investigation has been done into the correlation of thrombin generation and cardiac catheterization results in ischemic heart disease patients.

In the current research the investigator will investigate the correlation of thrombin generation values using calibrated automated thrombogram and cardiac catheterization results in active ischemic heart disease patients.

DETAILED DESCRIPTION:
The aim of our study is to investigate the correlation of thrombin generation values using calibrated automated thrombogram and cardiac catheterization results in active ischemic heart disease patients.

In total 340 patients are planned for inclusion in this trial. After signing an informed consent a blood sample will be obtained from each participant. the investigators will measure the thrombin generation over time in plasma assessed by the calibrated automated thrombogram (CAT). In addition information about the course and results of cardiac catheterization will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome: ST segment elevation myocardial infraction, unstable angina, non ST elevation myocardial infraction or patients presented with chest pain suspect for acute coronary syndrome .
* planned percutaneous coronary intervention.
* ability to give Informed consent.

Exclusion Criteria:

* Acute coronary syndrome in the last 6 month prior to current event.
* thrombophilia
* pregnancy
* liver failure or cirrhosis
* anticoagulant current use
* active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult with Acute coronary syndrome: ST segment elevation myocardial infraction, unstable angina, non ST elevation myocardial infraction or patients presented with chest pain suspect for acute coronary syndrome .
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
significant coronary lesion=>70% stenosis or =>50% stenosis in left main. | 1 week
  coronary arteries significant stenosis evaluated by percutaneous coronary intervention in ischemic heart disease patients
syntax score. | 1 week
  coronary arteries significant stenosis evaluated by percutaneous coronary intervention in ischemic heart disease patients

SECONDARY OUTCOMES:
The number of stenotic coronary arteries | 1 week
  the number of stenotic vessels in ischemic heart disease patients
Major adverse cardiac events (MACE) | 1 year
  MACE include acute coronary syndrome, cerebral vascular accident , revascularization, death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Elad, MD, Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- Hemek medical center, Afula, Israel